CLINICAL TRIAL: NCT07114510
Title: OPTImal Ventilation to Improve Pediatric Cardiac Arrest Outcomes (OPTI-VENT)
Brief Title: Optimal Ventilation for Cardiac Arrest
Acronym: OPTI-VENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Utah (Other); Villanova University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-022623; 1R01HD114622-01A1 (NIH)
Record Dates: First submitted 2025-07-31; First posted 2025-08-11 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Cardiac Arrest (CA)
Keywords: Pediatric
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Control (Experimental): Standard ICU resuscitation practices throughout study
  Interventions: Other: None - control
- OPTI-VENT Bundle (Experimental): Provider Education: During a brief (<2 minute) bedside education, the educator will 1) review the CPR ventilation rate targets for age, and 2) ensure the provider has a cue card of current rate recommendations on his/her person. Compliance will be defined as performance of at least 30 trainings per unit per month. We will record provider discipline and time since last training as a surrogate of training spread. Educators will leverage these two-minute trainings to review the patient's current ventilator settings as an initial target during CPR to ensure adequate chest rise.
  Additionally, a focus on CPR ventilation rates will be integrated into resuscitation education or quality meetings for all disciplines. "Report cards" detailing unit-level performance will be generated by the study team for review during site monthly presentations.
  Point-of-Care Guidance: A metronome will be deployed to all cardiac arrests using a smart phone application.
  Interventions: Other: OPTI-VENT Bundle
- Site 5 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 6 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 7 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 8 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 9 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 10 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 11 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 12 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 13 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 14 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 15 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control
- Site 16 (Experimental): Study enrollment will begin on the control arm. There will be a 2-month transition period as they onboard to the intervention. And the remainder of the study period will be on the OPTI-VENT Bundle intervention.
  Interventions: Other: OPTI-VENT Bundle; Other: Transition; Other: None - control

INTERVENTIONS:
Other: OPTI-VENT Bundle — Provider Education: During a brief (<2 minute) bedside education, the educator will 1) review the CPR ventilation rate targets for age, and 2) ensure the provider has a cue card of current rate recommendations on his/her person. Compliance will be defined as performance of at least 30 trainings per unit per month. We will record provider discipline and time since last training as a surrogate of training spread. Educators will leverage these two-minute trainings to review the patient's current ventilator settings as an initial target during CPR to ensure adequate chest rise.
  Additionally, a focus on CPR ventilation rates will be integrated into resuscitation education or quality meetings for all disciplines. "Report cards" detailing unit-level performance will be generated by the study team for review during site monthly presentations.
  Point-of-Care Guidance: A metronome will be deployed to all cardiac arrests using a smart phone application.
  Arms: OPTI-VENT Bundle; Site 10; Site 11; Site 12; Site 13; Site 14; Site 15; Site 16; Site 5; Site 6; Site 7; Site 8; Site 9
Other: Transition — There will be a 2-month transition period for study sites beginning study enrollment using standard ICU practices as they onboard to the study intervention.
  Arms: Site 10; Site 11; Site 12; Site 13; Site 14; Site 15; Site 16; Site 5; Site 6; Site 7; Site 8; Site 9
Other: None - control — Control - no intervention
  Arms: Control; Site 10; Site 11; Site 12; Site 13; Site 14; Site 15; Site 16; Site 5; Site 6; Site 7; Site 8; Site 9

SUMMARY:
Pediatric cardiac arrest is a life-threatening problem affecting >15,000 hospitalized children each year. Less than half of these children survive to hospital discharge, and neurologic morbidity is common among survivors. The objective of this study is to evaluate the effectiveness of the OPTI-VENT bundle to improve survival to discharge with favorable neurological outcome (Pediatric Cerebral Performance Category Score 1-2 or no change from baseline) among children receiving at least 1 minute of CPR.

ELIGIBILITY:
Inclusion Criteria:

* Invasive airway in place at the start of CPR or airway placed within the first 5 minutes
* Received at least 1 minute of CPR.

Exclusion Criteria:

* Lack of commitment to aggressive ICU therapies (e.g., CPR performed as part of end-of-life care.
* Brain death determination prior to the CPR event.
* Out-of-hospital cardiac arrest was the reason for initial admission to the hospital (known poor outcomes).
* Supported by Veno-Arterial Extra Corporeal Membrane Oxygenation at the start of CPR

Ages: 37 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1530 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Survival with a favorable neurologic outcome | From baseline (assessed prior to admission, or new in-hospital baseline assessed no more than 30 days prior to cardiac arrest for patients hospitalized >90 days) to the assessment at hospital discharge, estimated average of 6-12 months
  Survival to hospital discharge with a favorable neurologic outcome (Pediatric Cerebral Performance Category (PCPC) score (scored on a scale of 1-6) at hospital discharge of 1 (normal), 2 (mild disability) or no worse than baseline). Percentage of subjects in control vs. intervention will be compared.

SECONDARY OUTCOMES:
Ventilation rate | Two minutes after CPR start through end of CPR
  Intra-arrest ventilation rate between 18 - 32 breaths per minute. Ventilation rate will be calculated as an event average, excluding the first two minutes of the event. Percentage of events achieving target in control vs. intervention will be compared.

OTHER OUTCOMES:
Return of spontaneous circulation (ROSC) lasting >20 minutes | Duration of CPR event through 20 minutes after CPR
  Percentage of events achieving ROSC in control vs. intervention will be compared.
Return of circulation (via ROSC or eCPR) | Duration of CPR event through 20 minutes after CPR
  Percentage of events achieving return of circulation in control vs. intervention will be compared.
Survival to discharge | From cardiac arrest to hospital discharge, estimated average of 6-12 months
  Percentage of subjects surviving to discharge in control vs. intervention will be compared.
Survival with no new morbidity (change in Functional Status Score (FSS) from baseline of < 3 points) | From baseline (assessed prior to admission, or new in-hospital baseline assessed no more than 30 days prior to cardiac arrest for patients hospitalized >90 days) to the assessment at hospital discharge, estimated average of 6-12 months
  FSS is scored on a scale of 1-5 (lower number is better function) across 6 functional categories (mental status, sensory, communication, motor function, feeding, respiratory). Percentage of subjects surviving with no new morbidity in control vs. intervention will be compared.
Intra-arrest cerebral oxygen saturation | Duration of CPR event
  Intra-arrest cerebral oxygen saturation as a continuous variable will be compared between intervention and control.
Intra-arrest diastolic blood pressure (DBP) | Duration of CPR event
  Invasive arterial blood pressure (mmHg) as a continuous variable will be compared between intervention and control.
Intra-Arrest Diastolic Blood Pressure (DBP) Target | Duration of CPR
  Percentage of patients achieving DBP targets (>25mmHg in infants < 1 year of age; >30mmHg in older children) will be compared between control vs. intervention.
Hyperoxia (PaO2 >300 mmHg) | During the first 24 hours after return of circulation.
  Percentage of subjects in control vs. intervention will be compared.
Hypocarbia (PaCO2 <30 mmHg) | During the first 24 hours after return of circulation.
  Percentage of subjects in control vs. intervention will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sutton, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (20):
- United States (20):
  - CHOC, Orange, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Children's Hospital Colorado, Denver, Colorado
  - Nemours Children's Health, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Children's Health, Indianapolis, Indiana
  - Stead Family Children's Hospital, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Cohen Children's Medical Center, New Hyde Park, New York
  - UNC Children's Hospital, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Dell Children's Medical Center, Austin, Texas
  - Medical City Children's Hospital, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - Seattle Children's, Seattle, Washington
  - Children's Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
We plan to make a public use dataset available on the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH) at the conclusion of the study. The public use data set will contain a randomly generated subject identification number but will not contain any personal or site identifiers. The cleaned, item-level spreadsheet data for all variables will be shared openly. Final files used to generate specific analyses to answer the Specific Aims and related results will also be shared.
  All study documents will be made available along with the public use data set. The study protocol and statistical analysis plan will be shared publicly. To facilitate interpretation of the data, a data dictionary will be created, shared, and associated with the relevant datasets.

REFERENCES:
- [Background] Jacobs I, Nadkarni V, Bahr J, Berg RA, Billi JE, Bossaert L, Cassan P, Coovadia A, D'Este K, Finn J, Halperin H, Handley A, Herlitz J, Hickey R, Idris A, Kloeck W, Larkin GL, Mancini ME, Mason P, Mears G, Monsieurs K, Montgomery W, Morley P, Nichol G, Nolan J, Okada K, Perlman J, Shuster M, Steen PA, Sterz F, Tibballs J, Timerman S, Truitt T, Zideman D; International Liason Committee on Resusitation. Cardiac arrest and cardiopulmonary resuscitation outcome reports: update and simplification of the Utstein templates for resuscitation registries. A statement for healthcare professionals from a task force of the international liaison committee on resuscitation (American Heart Association, European Resuscitation Council, Australian Resuscitation Council, New Zealand Resuscitation Council, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa). Resuscitation. 2004 Dec;63(3):233-49. doi: 10.1016/j.resuscitation.2004.09.008. PMID 15582757
- [Background] Niles DE, Dewan M, Zebuhr C, Wolfe H, Bonafide CP, Sutton RM, DiLiberto MA, Boyle L, Napolitano N, Morgan RW, Stinson H, Leffelman J, Nishisaki A, Berg RA, Nadkarni VM. A pragmatic checklist to identify pediatric ICU patients at risk for cardiac arrest or code bell activation. Resuscitation. 2016 Feb;99:33-7. doi: 10.1016/j.resuscitation.2015.11.017. Epub 2015 Dec 17. PMID 26703460
- [Background] Pollack MM, Holubkov R, Glass P, Dean JM, Meert KL, Zimmerman J, Anand KJ, Carcillo J, Newth CJ, Harrison R, Willson DF, Nicholson C; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Functional Status Scale: new pediatric outcome measure. Pediatrics. 2009 Jul;124(1):e18-28. doi: 10.1542/peds.2008-1987. PMID 19564265
- [Background] Pollack MM, Holubkov R, Funai T, Clark A, Moler F, Shanley T, Meert K, Newth CJ, Carcillo J, Berger JT, Doctor A, Berg RA, Dalton H, Wessel DL, Harrison RE, Dean JM, Jenkins TL. Relationship between the functional status scale and the pediatric overall performance category and pediatric cerebral performance category scales. JAMA Pediatr. 2014 Jul;168(7):671-6. doi: 10.1001/jamapediatrics.2013.5316. PMID 24862461
- [Background] Del Castillo J, Lopez-Herce J, Matamoros M, Canadas S, Rodriguez-Calvo A, Cechetti C, Rodriguez-Nunez A, Alvarez AC; Iberoamerican Pediatric Cardiac Arrest Study Network RIBEPCI. Hyperoxia, hypocapnia and hypercapnia as outcome factors after cardiac arrest in children. Resuscitation. 2012 Dec;83(12):1456-61. doi: 10.1016/j.resuscitation.2012.07.019. Epub 2012 Jul 25. PMID 22841610
- [Background] Berg RA, Sutton RM, Reeder RW, Berger JT, Newth CJ, Carcillo JA, McQuillen PS, Meert KL, Yates AR, Harrison RE, Moler FW, Pollack MM, Carpenter TC, Wessel DL, Jenkins TL, Notterman DA, Holubkov R, Tamburro RF, Dean JM, Nadkarni VM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network (CPCCRN) PICqCPR (Pediatric Intensive Care Quality of Cardio-Pulmonary Resuscitation) Investigators. Association Between Diastolic Blood Pressure During Pediatric In-Hospital Cardiopulmonary Resuscitation and Survival. Circulation. 2018 Apr 24;137(17):1784-1795. doi: 10.1161/CIRCULATIONAHA.117.032270. Epub 2017 Dec 26. PMID 29279413
- [Background] Reeder RW, Girling A, Wolfe H, Holubkov R, Berg RA, Naim MY, Meert KL, Tilford B, Carcillo JA, Hamilton M, Bochkoris M, Hall M, Maa T, Yates AR, Sapru A, Kelly R, Federman M, Michael Dean J, McQuillen PS, Franzon D, Pollack MM, Siems A, Diddle J, Wessel DL, Mourani PM, Zebuhr C, Bishop R, Friess S, Burns C, Viteri S, Hehir DA, Whitney Coleman R, Jenkins TL, Notterman DA, Tamburro RF, Sutton RM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network (CPCCRN). Improving outcomes after pediatric cardiac arrest - the ICU-Resuscitation Project: study protocol for a randomized controlled trial. Trials. 2018 Apr 3;19(1):213. doi: 10.1186/s13063-018-2590-y. PMID 29615134
- [Background] ICU-RESUS and Eunice Kennedy Shriver National Institute of Child Health; Human Development Collaborative Pediatric Critical Care Research Network Investigator Groups; Sutton RM, Wolfe HA, Reeder RW, Ahmed T, Bishop R, Bochkoris M, Burns C, Diddle JW, Federman M, Fernandez R, Franzon D, Frazier AH, Friess SH, Graham K, Hehir D, Horvat CM, Huard LL, Landis WP, Maa T, Manga A, Morgan RW, Nadkarni VM, Naim MY, Palmer CA, Schneiter C, Sharron MP, Siems A, Srivastava N, Tabbutt S, Tilford B, Viteri S, Berg RA, Bell MJ, Carcillo JA, Carpenter TC, Dean JM, Fink EL, Hall M, McQuillen PS, Meert KL, Mourani PM, Notterman D, Pollack MM, Sapru A, Wessel D, Yates AR, Zuppa AF. Effect of Physiologic Point-of-Care Cardiopulmonary Resuscitation Training on Survival With Favorable Neurologic Outcome in Cardiac Arrest in Pediatric ICUs: A Randomized Clinical Trial. JAMA. 2022 Mar 8;327(10):934-945. doi: 10.1001/jama.2022.1738. PMID 35258533
- [Background] Aufderheide TP, Sigurdsson G, Pirrallo RG, Yannopoulos D, McKnite S, von Briesen C, Sparks CW, Conrad CJ, Provo TA, Lurie KG. Hyperventilation-induced hypotension during cardiopulmonary resuscitation. Circulation. 2004 Apr 27;109(16):1960-5. doi: 10.1161/01.CIR.0000126594.79136.61. Epub 2004 Apr 5. PMID 15066941
- [Background] Aufderheide TP, Lurie KG. Death by hyperventilation: a common and life-threatening problem during cardiopulmonary resuscitation. Crit Care Med. 2004 Sep;32(9 Suppl):S345-51. doi: 10.1097/01.ccm.0000134335.46859.09. PMID 15508657
- [Background] Grieco DL, J Brochard L, Drouet A, Telias I, Delisle S, Bronchti G, Ricard C, Rigollot M, Badat B, Ouellet P, Charbonney E, Mancebo J, Mercat A, Savary D, Richard JM. Intrathoracic Airway Closure Impacts CO2 Signal and Delivered Ventilation during Cardiopulmonary Resuscitation. Am J Respir Crit Care Med. 2019 Mar 15;199(6):728-737. doi: 10.1164/rccm.201806-1111OC. PMID 30257100
- [Background] Chapman JD, Geneslaw AS, Babineau J, Sen AI. Improving Ventilation Rates During Pediatric Cardiopulmonary Resuscitation. Pediatrics. 2022 Sep 1;150(3):e2021053030. doi: 10.1542/peds.2021-053030. PMID 36000325
- [Background] Sutton RM, Niles D, Meaney PA, Aplenc R, French B, Abella BS, Lengetti EL, Berg RA, Helfaer MA, Nadkarni V. Low-dose, high-frequency CPR training improves skill retention of in-hospital pediatric providers. Pediatrics. 2011 Jul;128(1):e145-51. doi: 10.1542/peds.2010-2105. Epub 2011 Jun 6. PMID 21646262
- [Background] Sutton RM, Reeder RW, Landis WP, Meert KL, Yates AR, Morgan RW, Berger JT, Newth CJ, Carcillo JA, McQuillen PS, Harrison RE, Moler FW, Pollack MM, Carpenter TC, Notterman DA, Holubkov R, Dean JM, Nadkarni VM, Berg RA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network (CPCCRN). Ventilation Rates and Pediatric In-Hospital Cardiac Arrest Survival Outcomes. Crit Care Med. 2019 Nov;47(11):1627-1636. doi: 10.1097/CCM.0000000000003898. PMID 31369424
- [Background] Topjian AA, Raymond TT, Atkins D, Chan M, Duff JP, Joyner BL Jr, Lasa JJ, Lavonas EJ, Levy A, Mahgoub M, Meckler GD, Roberts KE, Sutton RM, Schexnayder SM; Pediatric Basic and Advanced Life Support Collaborators. Part 4: Pediatric Basic and Advanced Life Support: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S469-S523. doi: 10.1161/CIR.0000000000000901. Epub 2020 Oct 21. No abstract available. PMID 33081526
- [Background] Nadkarni VM, Larkin GL, Peberdy MA, Carey SM, Kaye W, Mancini ME, Nichol G, Lane-Truitt T, Potts J, Ornato JP, Berg RA; National Registry of Cardiopulmonary Resuscitation Investigators. First documented rhythm and clinical outcome from in-hospital cardiac arrest among children and adults. JAMA. 2006 Jan 4;295(1):50-7. doi: 10.1001/jama.295.1.50. PMID 16391216
- [Background] Wolfe H, Zebuhr C, Topjian AA, Nishisaki A, Niles DE, Meaney PA, Boyle L, Giordano RT, Davis D, Priestley M, Apkon M, Berg RA, Nadkarni VM, Sutton RM. Interdisciplinary ICU cardiac arrest debriefing improves survival outcomes*. Crit Care Med. 2014 Jul;42(7):1688-95. doi: 10.1097/CCM.0000000000000327. PMID 24717462
- [Background] Girotra S, Nallamothu BK, Spertus JA, Li Y, Krumholz HM, Chan PS; American Heart Association Get with the Guidelines-Resuscitation Investigators. Trends in survival after in-hospital cardiac arrest. N Engl J Med. 2012 Nov 15;367(20):1912-20. doi: 10.1056/NEJMoa1109148. PMID 23150959
- [Background] Holmberg MJ, Ross CE, Fitzmaurice GM, Chan PS, Duval-Arnould J, Grossestreuer AV, Yankama T, Donnino MW, Andersen LW; American Heart Association's Get With The Guidelines-Resuscitation Investigators. Annual Incidence of Adult and Pediatric In-Hospital Cardiac Arrest in the United States. Circ Cardiovasc Qual Outcomes. 2019 Jul 9;12(7):e005580. PMID 31545574

DOCUMENTS (1):
  • Study Protocol (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT07114510/Prot_000.pdf